CLINICAL TRIAL: NCT03645291
Title: Comparison of Skin Prick Testing and Intradermal Skin Test Result of Local and Imported Insect Allergen Extracts in Patients With Severe Insect Sting Allergy
Brief Title: Comparison of Skin Prick Testing and Intradermal Skin Test Result of Local and Imported Insect Allergen Extracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 450/2559 (EC 3)
Record Dates: First submitted 2018-08-16; First posted 2018-08-24 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Allergy to Arthropod Sting
Keywords: insect sting allergy; Hymenoptera allergy; local insect allergen extracts
MeSH Terms: conditions — Venom Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Comparison of skin prick testing and Intradermal skin test result of local and imported insect allergen extracts in patients with severe insect sting allergy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: None of the patients and participants know the type of insect allergen extracts used in skin prick and intradermal test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin test with local extract (Active Comparator): Skin prick test and intradermal test with local stinging insect allergen extracts that develop in Immunological division of Siriraj hospital, mahidol University
  Interventions: Diagnostic Test: Local insect allergen extracts skin test
- Skin test with commercial extract (Sham Comparator): Skin prick test and intradermal test with commercial stinging insect allergen extracts that order from ALK company
  Interventions: Diagnostic Test: Local insect allergen extracts skin test

INTERVENTIONS:
Diagnostic Test: Local insect allergen extracts skin test — Every patient received both local and commercial insect allergen extracts but in blinded methods
  Other Names: commercial insect allergen extracts from ALK skintest

SUMMARY:
Comparison the results of skin prick testing and Intradermal skin test result of local and imported insect allergen extracts in patients with serious insect sting allergy reactions

DETAILED DESCRIPTION:
The patients with serious insect sting allergy reactions were evaluated and skin prick test and intradermal test with local and imported insect allergen extracts were performed. Specific IgE for insects was also performed. The results of skin prick testing and Intradermal skin test of local and imported insect allergen extracts were compared. The results also compared with specific IgE to insects

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe insect allergy reaction
* Allow being done skin test and blood foe specific IgE

Exclusion Criteria:

* Serious systemic diseases
* severe asthma
* pregnant or nursing
* severe and extended skin lesion

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Comparison of positive skin test results of local and commercial insect allergen extracts | 1 year
  Measure wheal size of skin test of local and commercial insect allergen extracts then compare the positive result and wheal size between local and commercial extracts.

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Publication